CLINICAL TRIAL: NCT05407701
Title: Countermeasure Influence of 4-Weeks Cranberry Ingestion on Immune Dysfunction, Inflammation, and Muscle Damage Induced by Intensive Cycling
Brief Title: Cranberry Ingestion and Cycling Related Immunity and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-0114
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Response; Metabolic Disturbance; Immune Suppression
Keywords: Cranberries; exercise; immune function; oxylipins; proteomics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized treatment, double blinded procedures, crossover
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation, with the cranberry and placebo beverages of the same taste and color, and contained in identical looking bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry (Experimental): 100% juice active: water, cranberry juice concentrate.
  Interventions: Dietary Supplement: Cranberry Juice
- Placebo (Placebo Comparator): 100% juice placebo: water, fructose, dextrose, citric acid, malic acid, natural flavors, pectin, cherry colorant, sucralose.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry Juice — 100% cranberry juice
  Arms: Cranberry
Dietary Supplement: Placebo — Placebo juice
  Arms: Placebo

SUMMARY:
This is a randomized, crossover clinical trial with 25 male and female cyclists. Study participants will ingest polyphenol-rich cranberry juice or placebo juice for 4 weeks under double-blinded procedures, and then crossover to the opposite supplement. The primary objective of this study is to examine the efficacy of 4-weeks ingestion of cranberry juice in moderating exercise-induced inflammation, immune dysfunction, and muscle damage. Outcome measures will include global proteiomics, oxylipins, and cytokines.

DETAILED DESCRIPTION:
RESEARCH DESIGN: Subjects will come to the lab for orientation/baseline testing, pre-and post-supplementation (4 weeks cranberry ingestion compared to water alone) blood, stool, and urine sample collections with 3-d food records, two 2.25 h cycling sessions, and additional lab visits to provide 1-day 7:00 am recovery blood and saliva samples) (thus 7 total lab visits). The total amount of time subjects will be asked to volunteer for this study is about 16 hours at the Human Performance Laboratory (over a 10-week period).

1.A. Orientation/Baseline Testing (Visit #1) After voluntarily signed IRB-approved consent forms, study participants will be tested for maximal aerobic capacity (VO2max) during a graded, cycling test with continuous metabolic monitoring with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Demographic and training histories will be acquired with questionnaires. 3-day food records, 24-h urine collection kits, and stool collection kits will be supplied with thorough instructions.

B. Pre-Supplementation Lab Visit #2 and 4-Week Cranberry Supplementation Protocol: Four weeks prior to the first cycling session, subjects will report to the Human Performance Laboratory at approximately 7:00-8:00 am. DOMS and POMS questionnaires will be administered. To assess potential adverse effects, a symptom inventory will be conducted using a 4-week retrospective questionnaire (before and after the 4-week supplementation period). Blood and saliva samples will be collected in an overnight fasted state to coincide with the same time of the day for the post-supplementation blood draw. Urine samples, stool samples, and 3-d food records will be turned in. A 4-week supply of cranberry juice or placebo will be given to the participants, with instructions to consume 4 fl. Oz. each with the first and last meals of the day (8 fl. Oz. per day for 4 weeks). Subjects will be instructed to store and then bring the cranberry and placebo beverage containers to their next lab visit (to verify compliance). Subjects will be given a 10-week log book to record daily whether or not they are sick and the severity of their symptoms.

C. 2.25 h Cycling Session (Lab Visit #3): During the 3-day period prior to the 2.25-h cycling session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, and polyphenols. Subjects will record all food and beverage intake during the 3-day period, with macro- and micro-nutrient intake assessed using the Food Processor dietary analysis software system (ESHA Research, Salem, OR). We will also measure total flavonoid intake (and 6 flavonoid subgroups) using the USDA flavonoid database that we have incorporated into the Food Processor database (9). Study participants will report to the Human Performance Lab in an overnight fasted state, turn in urine and stool samples, provide blood and saliva samples, ingest 1 cup cranberry with 1 cup of water, or 1 cup of water alone, and then cycle 2.25 h at high intensity (70% VO2max) while ingesting water alone (3 ml/kg every 15 minutes). A sweat patch will be applied to the lower back before exercise begins and then taken off immediately after the exercise bout is complete (https://www.epicorebiosystems.com/gx-sweat-patch/). Blood and saliva samples will be collected at 0 h, 1.5 h, 3.0 h, and 24 h post-exercise.

Testing protocol during the lab sessions with the 2.25-h run session:

1. 7:00 am: Provide blood and saliva samples, delayed onset of muscle soreness (DOMS) rating (1-10 scale), profile of mood states ratings (POMS), and turn in the 24-h urine sample, stool sample, and 3-day food record. Fill in the 4-week retrospective symptom log.
2. 7:10 am: Ingest 4 fl. Oz. cranberry or 4 fl. Oz. placebo. A sweat patch will be applied to the lower back.
3. 7:30 am: Start the 2.25 h cycling session. Subjects will cycle on lab trainers at 70% VO2max (~marathon race pace) for 2.25 hours. Oxygen consumption, carbon dioxide production, respiratory exchange ratio, and ventilation will be measured using the Cosmed Quark CPET metabolic cart after 15 minutes and then every 30 minutes. Subjects will consume 3 ml/kg water every 15 min. No other beverage or food containing energy or nutrients will be allowed during the 2.25-h cycling sessions.
4. ~10:00 am to 1:00 pm: The sweat patch will be removed. Blood and saliva samples will be taken via venipuncture immediately after completing the cycling session, and then 1.5-h and 3.0-h post-exercise. Subjects will be allowed to shower and change clothes. The DOMS and POMS questionnaires will be administered each time blood and saliva samples are collected. Subjects will ingest no food or beverage other than water (7 ml/kg during the 1.5 h post-exercise period). After the 1.5 h post-exercise blood draw, subjects will consume Boost (8 kcal per kilogram of body weight). Another blood sample will be collected 3-h post-exercise. Afterwards, subjects will be allowed to leave the lab with instructions to adhere to the food list requirements, and to keep exercise training moderate.
5. 7:00 am, next morning: 24-h blood sample and DOMS and POMS ratings (Lab visit #4).

D. Washout/Crossover/Repeat Subjects will engage in a 4-week washout period without the cranberry supplements, crossover to the opposite treatment arm, and then repeat all procedures (Lab visits #5,6,7).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cyclist, ages 18-55 years, and capable of cycling 2.25 h in the lab on trainers at 70% VO2max (close to race pace).
* Non-smoker
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation (especially NSAIDs) for the duration of the 10-week study.
* Agree to taper their exercise routine prior to each of the two lab cycling sessions.
* Agree to avoid ingestion of cranberry products during the study (other than provided).

Exclusion Criteria:

* Inability to comply with study requirements.
* History of allergic reactions to cranberry ingestion.
* Females: body weight below 110 pounds; pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the principle investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Blood lymphocyte proliferation | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  The mitogenic response of lymphocytes will be determined in whole blood culture using suboptimal mitogen (Concanavalin A) doses

SECONDARY OUTCOMES:
Plasma lipid mediators | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of arachadonic acid oxidized derivatives from LC-MS-MS analysis
Plasma proteins | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of immune- and inflammation-related proteins from proteomics profiling using LC-MS-MS analysis
Plasma cytokine panel | Change from pre-study to post-4 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of cytokines most influenced by exercise inclduing IL6, IL8, IL10, MCP-1, IL1ra, GCSF

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December, 2022, indefinitely
Access Criteria: Upon request